CLINICAL TRIAL: NCT07131085
Title: Clinical Study on the Safety and Efficacy of QH101 in Patients With Relapsed/Refractory Acute Myeloid Leukemia(R/R AML) and Relapsed/Refractory Myelodysplastic Syndromes(R/R MDS)
Brief Title: QH101 Cell Therapy Relapsed/Refractory(R/R) Acute Myeloid Leukemia(AML) and Myelodysplastic Syndromes(MDS)
Status: Not yet recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Anhui Provincial Hospital (Other Government)
Responsible Party: Principal Investigator, Xiaoyu Zhu, Director of Hematology Department, Anhui Provincial Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: QH10104-RML-01（0）
Record Dates: First submitted 2025-08-05; First posted 2025-08-20 (Actual); Last update posted 2025-08-20 (Actual); Status verified 2025-08

CONDITIONS: MDS; AML
Keywords: TCR; BTN; γδT; allogeneic; cell therapy
MeSH Terms: interventions — fludarabine; Cyclophosphamide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Patients with R/R AML or MDS (Experimental): Patients with R/R AML or MDS. A conditioning chemotherapy regimen of fludarabine and cyclophosphamide will be administered followed by investigational treatment, QH101 product.
  Interventions: Drug: Allogeneic TCR-enhanced γδ T cell(QH101); Drug: Fludarabine (FLU); Drug: Cyclophosphamide (CTX)

INTERVENTIONS:
Drug: Allogeneic TCR-enhanced γδ T cell(QH101) — dose escalation (3+3) : dose 1 (5×10^8 enTCR γδ cells) , dose 2 (1.5×10^9 enTCR γδ cells), dose 3 (3×10^9 enTCR γδ cells)
Drug: Fludarabine (FLU) — Intravenous fludarabine 20~30 mg/m^2/day on days -5, -4, and -3
Drug: Cyclophosphamide (CTX) — Intravenous cyclophosphamide 300~500 mg/m^2/day on days -5, -4, and -3.

SUMMARY:
QH101 is an allogeneic TCR-enhanced Vδ2 T cell therapy product engineered to express BTN protein-specific binding elements on the cell surface. This innovative approach harnesses the natural cytotoxic capabilities of Vδ2 T cells while augmenting their ability to recognize BTN proteins, thereby significantly improving tumor cell elimination efficiency. Notably, QH101 is designed without co-stimulatory signal domains or the CD3ζ domain, which prevents T cell exhaustion from overactivation and effectively enhances in vivo persistence.

Patients with R/R AML face particularly poor prognoses, with conventional chemotherapy and targeted therapies achieving suboptimal complete remission rates and long-term survival below 10%. Similarly, R/R MDS patients typically demonstrate median overall survival of less than one year (with TP53-mutated cases showing even poorer outcomes of 3-6 months), making clinical trial participation the most viable therapeutic option.

The development of effective treatments for R/R AML/MDS presents significant challenges due to:1)The paucity of disease-specific molecular targets;2)The slow progress in drug development. Allogeneic γδ T-cell therapy featuring enhanced TCR functionality and multi-mechanism tumoricidal activity represents a promising investigational approach for addressing R/R AMLMDS. This innovative strategy combines the advantages of: 1)Improved target recognition through TCR enhancement; 2)Multi-faceted tumor-killing mechanisms; 3)Potential for better safety and persistence profiles.

ELIGIBILITY:
Selection criteria:

1. Age ≥ 14 years, no gender restrictions;
2. Diagnosed with AML according to the standards of the NCCN (2024 V2), ELN (2023), and the Chinese "Guidelines for the Diagnosis and Treatment of AML (2024 Edition)"; or diagnosed with MDS according to the standards of the NCCN (2024 V2), ELN (2023), and the Chinese "Expert Consensus on the Diagnosis and Treatment of MDS (2024 Edition)"; （1） Meets the criteria for R/R AML, including any of the following:

   1. Relapsed: Leukemic cells reappear in the peripheral blood after complete remission, or Leukemic blasts≥5% in the bone marrow (excluding other causes such as bone marrow regeneration after consolidation chemotherapy), or leukemic cell infiltration in extramedullary sites;
   2. Refractory: Primary cases that fail to respond to two cycles of standard treatment, or cases that relapse within 12 months after consolidation intensive therapy following complete remission (CR), or cases that relapse after 12 months and fail to respond to conventional chemotherapy, or cases with two or more relapses, or cases with persistent extramedullary leukemia; （2）Meets the criteria for R/R MDS, including any of the following conditions:

   <!-- -->

   1. Relapsed: Patients who have achieved hematologic improvement or CR but subsequently experience hematologic decline (e.g., hemoglobin <10 g/dL, platelets <50×10⁹/L, neutrophils <1.0×10⁹/L), or an increase in the proportion of blast cells in the bone marrow (≥5%), or the emergence of new cytogenetic abnormalities or molecular progression (e.g., increased TP53 mutation burden);
   2. Refractory: No hematologic or bone marrow improvement after ≥4-6 cycles of hypomethylating agent (HMA) therapy (e.g., azacitidine or decitabine), or low-risk MDS resistant to erythropoietin or immunomodulatory agents (e.g., lenalidomide).
3. Expected survival time exceeds 3 months;
4. Eastern Cooperative Oncology Group (ECOG) performance status is 0-2;
5. Organ function meets the following requirements: 1)Liver function must meet: ALT ≤ 3 × ULN; AST ≤ 3 × ULN; Total bilirubin ≤ 3.0 × ULN. 2)Renal function must meet the following criteria: Serum creatinine ≤ 1.5 × upper limit of normal (ULN); 3)Cardiac function: Echocardiogram showing left ventricular ejection fraction ≥ 50%; 4)Pulmonary function: Normal oxygen saturation without oxygen supplementation.
6. Female participants of childbearing potential and male participants whose partners are of childbearing potential must use medically approved contraceptive measures or abstain from sexual intercourse during the study treatment period and for at least 6 months after the study treatment period. Female participants of childbearing potential must have a negative serum HCG test within 7 days prior to study enrollment and must not be breastfeeding.
7. No significant genetic disorders;
8. The subject or their legal guardian voluntarily participates in this study, understands the trial information, objectives, and risks described in the informed consent form, and can provide a signed and dated informed consent form;
9. The subject or their legal guardian is willing and able to comply with all trial requirements.

Exclusion criteria:

1. Patients with a history of severe central nervous system disorders, such as uncontrolled epileptic seizures, stroke, severe brain injury with aphasia, paralysis, dementia, Parkinson's disease, or mental disorders;
2. New York Heart Association (NYHA) Class III or IV heart failure;
3. Undergone coronary angioplasty, coronary stent implantation, or coronary artery bypass surgery; or experienced thrombotic or embolic events (e.g., cerebrovascular events [including transient ischemic attacks, but excluding lacunar cerebral infarction], deep vein thrombosis [excluding deep vein thrombosis caused by PICC catheter placement], pulmonary embolism, etc.);
4. Presence of disseminated intravascular coagulation;
5. Presence of severe autoimmune diseases or immunodeficiency disorders;
6. Presence of active graft-versus-host disease requiring ongoing systemic treatment;
7. Subjects currently receiving systemic steroid or other immunosuppressive therapy prior to screening, and who are determined by the investigator to require long-term use of such therapy after enrollment (excluding inhaled or topical use);
8. Other severe medical conditions deemed inappropriate for enrollment by the investigator (e.g., uncontrolled hypertension or diabetes, severe renal insufficiency, severe pulmonary dysfunction, etc.);
9. Active HBV or HCV infection (HBV-DNA positive or HCV-RNA positive), HIV-positive, or positive syphilis test results;
10. Other severe or persistent active infections;
11. Adverse events related to systemic immunotherapy (including other investigational drugs or medical device interventions) prior to screening have not yet decreased to Grade 1 severity or returned to baseline status;
12. Discontinuation of immunosuppressive agents for less than 2 weeks;
13. History of allergy to any component of the cellular product;
14. Vaccination or any surgical procedure within 4 weeks prior to screening;
15. Other conditions deemed by the investigator to potentially increase the risk to the subject or interfere with trial results.

Min Age: 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 9 (Estimated)
Dates: Start 2025-08-15 (Estimated); Primary Completion 2027-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Incidence of AE | 12 months
  AE is defined as any adverse medical event occurring from the date of lymphocyte depletion to 12 months after QH101 infusion. Among these, cytokine release syndrome (CRS) and immune cell-associated neurotoxicity syndrome (ICANS) are graded according to the standards set by the American Society for Transplantation and Cellular Therapy (ASTCT). Graft-versus-host disease (GVHD) is graded according to the standards defined by the Mount Sinai Acute GVHD International Consortium. Other AEs are graded according to the Common Terminology Criteria for Adverse Events (CTCAE) v5.0.
Incidence of dose-limiting toxicity (DLT) | Within 28 days post-cell infusion

SECONDARY OUTCOMES:
Pharmacokinetics: Persistence of QH101 | 12 months
  Persistence of QH101 assessed by number in peripheral blood.
Overall response rate (ORR) | 12 months
  The proportion of subjects achieving CR (complete remission)/CRh (complete remission with partial hematological recovery)/CRi (complete remission with incomplete hematological recovery)/PR (partial remission)
Immunogenicity: Proportion of subjects with anti drug antibody (ADA) | 12 months
Pharmacodynamics: Peak level of cytokines in serum | Up to 28 days after infusion
  The cytokines mainly include interleukin-2 (IL-2 ), IL-6, IL-8, IL-10, tumor necrosis factor-α (TNF-α), interferon-γ(IFN-γ). Peak was defined as the maximum post-baseline level of the cytokine.